CLINICAL TRIAL: NCT04855890
Title: HIgh Power Short Duration Radiofrequency Ablation or Cryoballoon Ablation for Paroxysmal Atrial Fibrillation - the HIPAF Trial
Brief Title: HIgh Power Short Duration Radiofrequency Ablation or Cryoballoon Ablation for Paroxysmal Atrial Fibrillation
Acronym: HIPAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Köln (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIPAF-21
Record Dates: First submitted 2021-04-20; First posted 2021-04-22 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Atrial Fibrillation and Flutter; Atrial Fibrillation; Paroxysmal Atrial Fibrillation
Keywords: atrial fibrillation; high power short duration; pulmonary vein isolation; cryo-ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: The present study is a mono-center prospective randomized study enrolling 170 patients with PAF and no prior Ablation for AF.
  Patients will be randomized to one of the following groups. Group A: Cryo-Ablation PVI will be performed using a Cryo-balloon. Group B: High-Power-Short-Duration PVI will be performed using HPSD RF-ablation. (70W over 5s posterior and 7s anterior) Catheter ablation procedures will be performed with commercially available devices including 3D mapping systems (EnSite, Abbott) and irrigated radiofrequency current (RFC) ablation or cryothermal balloon ablation (Arctic Front Advance Pro, Medtronic).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryo-Ablation (Active Comparator): Cryo-Balloon (Arctic Front Advance ProTM, Medtronic, Minneapolis, MN, USA) will be advanced to the LA and navigated to the PV's using an inner-lumen circular mapping catheter (Achieve AdvanceTM, Medtronic, Minneapolis, MN, USA). After confirming complete PV sealing by the CB using occlusion angiograms cryothermal energy will be applied for min 120 seconds aiming at PV isolation of all PV's according to the clinical standard.
  Interventions: Procedure: Ablation
- High Power Short Duration-Ablation (Active Comparator): A detailed electroanatomical map of the left atrium during sinus rhythm will be acquired using Ensite (Abbott, St. Paul, MN, USA).
  Upon completion of the LA map, a second transseptal puncture will be performed in order to insert an ablation catheter. To achieve antral PVI irrigated radiofrequency current ablation will be performed using a power of 70W and a flush rate of 8-30ml/min with a duration of 5 seconds for the anterior and 7 seconds for the posterior LA. Ablation catheters used will contain Flexibilty (Abbott, St. Paul, MN, USA) and TactiFlex (Abbott, St. Paul, MN, USA).
  Interventions: Procedure: Ablation

INTERVENTIONS:
Procedure: Ablation — The ablation procedure will be performed during deep sedation using midazolam, fentanyl and a continuous infusion of propofol. Vital parameters will be monitored. For catheter access three 8F sheaths will be inserted into the femoral veins. A multipolar diagnostic catheter will be placed in the coronary sinus. Single transseptal puncture and insertion of a 8.5 F transseptal sheath or 12F Cryo-Sheath (FlexCath AdvanceTM, Medtronic, Minneapolis, MN, USA) will be followed by PV angiographies. Before or shortly after transseptal puncture unfractionated heparin will be repeatedly administered to maintain an activated clotting time between 250 and 400s.

SUMMARY:
Pulmonary vein isolation (PVI) using the cryoballoon has been proven equal to RF-PVI and is widely used. High Power Short Duration Ablation in RF-PVI has been successfully tested in several trials. Prospective data comparing both strategies is lacking.

This trial will compare acute success rates, safety and foremost long-term outcome of two different PVI strategies (HPSD-PVI vs. cryo-PVI).

DETAILED DESCRIPTION:
In several trials and real-life data pulmonary vein isolation (PVI) using the cryoballoon technique has been proven equal to RF-PVI for the treatment of paroxysmal atrial fibrillation (PAF). Due to the "single-shot character" of the device and shorter procedure times the cryoballoon is being widely used for PVI within the last years. However, additional endpoints such as "non-excitability" of the ablation line and consecutive arrhythmias may not be targeted properly by this device also lacking a detailed contact map to evaluate potential fibrotic areas.

For the past decade, the use of RF energy for successful PVI has been the "gold standard". However, ablation time and potential gaps within the circumferential ablation line are still an issue. High power (70 Watts) over short duration (7s) (HPSD) is a recently introduced RF-PVI concept. It has been shown to be as effective as conventional RF-PVI with equal safety features, shorter procedure durations and a superior long-term outcome. Therefore, HPSD-PVI in combination with the endpoint of "non-excitability" is potentially superior with regard to freedom of atrial arrhythmia during long-term FU compared to cryo-PVI with similar procedure times.

So far, randomized prospective data comparing HPSD versus cryo-PVI are lacking.

The aim of this prospective randomized study is to compare acute success rates, safety and foremost long-term outcome of two different PVI strategies (HPSD-PVI vs. cryo-PVI):

1. To find the safest and most effective treatment strategy for PAF patients. 2. To evaluate the risk of complications for both treatment strategies.

3. Evaluation of procedure endpoints like duration, costs and radiation dose.

The present study is a mono-center prospective randomized study enrolling 170 patients with PAF and no prior Ablation for AF.

Patients will be randomized to one of the following groups. Group A: Cryo-Ablation PVI will be performed using a Cryo-balloon. Group B: High-Power-Short-Duration PVI will be performed using HPSD RF-ablation. (70W over 5s posterior and 7s anterior) Catheter ablation procedures will be performed with commercially available devices including 3D mapping systems (EnSite, Abbott) and irrigated radiofrequency current (RFC) ablation or cryothermal balloon ablation (Arctic Front Advance Pro, Medtronic).

The study shall start enrolling patients in April 2021. The last patient shall be enrolled in January 2023. Since follow-up is 12 months, end of study is planned for January 2024.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic non-valvular atrial fibrillation with no prior ablation with an indication for re-ablation according to current guidelines.
* Age 18-85 years.
* Patient is able to provide informed consent and is willing to comply with the study protocol.

Exclusion Criteria:

* Contraindications for left atrial ablation
* History of interventional or surgical AF-ablation
* History of stroke during the past 12 months
* BMI >40kg/m2
* History of mitral valve surgery
* Severe mitral valve regurgitation
* Inability to be treated with oral anticoagulation
* Presence of intracardiac thrombi
* Contraindication or absolute indication for one of the two strategies
* Pregnancy
* Participation in other clinical studies
* Unwilling to follow the study protocol and to attend follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence of atrial arrhythmia | 12 months after a 3 months blanking period
  Combined primary endpoint of recurrent atrial arrhythmia, onset of new AAD or re- ablation of atrial arrhythmia during the follow-up of 12 months after a 3-months blanking period.

SECONDARY OUTCOMES:
Periprocedural complications | Within 48 hours of procedure
  Incidence of peri-procedural complications such as: major bleeding requiring intervention, phrenic nerve palsy, pericardial tamponade, thrombembolic events, death.
Number of re-hospitalisations | 12 months after a 3 months blanking period
  Number of re-hospitalisations (total and for cardiovascular reasons)
Cardioversions | 12 months after a 3 months blanking period
  Number of electrical cardioversions
Procedural data | During the procedure
  Procedure duration, radiation dose, radiation duration

CONTACTS AND LOCATIONS:
Overall Officials: Arian Sultan, PD Dr., Principal Investigator — University of Cologne, Heart Center, Dept. of Electrophysiology; Daniel Steven, Prof. Dr., Principal Investigator — University of Cologne, Heart Center, Dept. of Electrophysiology
Locations (1):
- Department of electrophysiology, Heart Center Cologne, University of Cologne, Cologne, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirchhof P, Benussi S, Kotecha D, Ahlsson A, Atar D, Casadei B, Castella M, Diener HC, Heidbuchel H, Hendriks J, Hindricks G, Manolis AS, Oldgren J, Popescu BA, Schotten U, Van Putte B, Vardas P; ESC Scientific Document Group. 2016 ESC Guidelines for the management of atrial fibrillation developed in collaboration with EACTS. Eur Heart J. 2016 Oct 7;37(38):2893-2962. doi: 10.1093/eurheartj/ehw210. Epub 2016 Aug 27. No abstract available. PMID 27567408
- [Background] Kuck KH, Brugada J, Furnkranz A, Metzner A, Ouyang F, Chun KR, Elvan A, Arentz T, Bestehorn K, Pocock SJ, Albenque JP, Tondo C; FIRE AND ICE Investigators. Cryoballoon or Radiofrequency Ablation for Paroxysmal Atrial Fibrillation. N Engl J Med. 2016 Jun 9;374(23):2235-45. doi: 10.1056/NEJMoa1602014. Epub 2016 Apr 4. PMID 27042964
- [Background] Murray MI, Arnold A, Younis M, Varghese S, Zeiher AM. Cryoballoon versus radiofrequency ablation for paroxysmal atrial fibrillation: a meta-analysis of randomized controlled trials. Clin Res Cardiol. 2018 Aug;107(8):658-669. doi: 10.1007/s00392-018-1232-4. Epub 2018 Mar 21. PMID 29564527
- [Background] Kottmaier M, Popa M, Bourier F, Reents T, Cifuentes J, Semmler V, Telishevska M, Otgonbayar U, Koch-Buttner K, Lennerz C, Bartkowiak M, Kornmayer M, Rousseva E, Brkic A, Grebmer C, Kolb C, Hessling G, Deisenhofer I. Safety and outcome of very high-power short-duration ablation using 70 W for pulmonary vein isolation in patients with paroxysmal atrial fibrillation. Europace. 2020 Mar 1;22(3):388-393. doi: 10.1093/europace/euz342. PMID 31872249